CLINICAL TRIAL: NCT01240317
Title: eVENT: An Expert System for Detecting Critical Events During Anesthesia (Human Patient Simulator Study)
Brief Title: eVent in the Human Patient Simulator
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Mark Ansermino, Principle Investigator, University of British Columbia
Other Study IDs: H10-02621
Record Dates: First submitted 2010-11-10; First posted 2010-11-15 (Estimated); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Efficacy of the Expert System's Ability to Help Detect Critical Events
Keywords: expert system; decision support system; human patient simulator; anesthesia

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
In this study, the investigators are testing the expert system called eVENT. eVENT provides expert advice about the patient's breathing. The investigators have developed and tested a prototype of eVENT and now want to test how it works in practice. To do this the investigators plan to use computer based simulations and test it when used by anesthesiologists in a full size human simulator. If these tests are successful the investigators will then be ready to evaluate eVENT on real patients.

DETAILED DESCRIPTION:
The development of new sensors or the intelligent synthesis of existing signals (smart sensors) cannot reliably prevent adverse events unless the investigators assimilate the data produced from these devices and provide it to the clinician in a format that is easy to comprehend. The expert system that the investigators are developing will provide intelligent synthesis of data. The clinician focus can then be directed toward the patient rather than continual observation of the monitors.

Clinicians need an expert system to augment vigilance and situation awareness, and to aid in decision making to prevent patient harm.

The development of an expert system to assist the everyday anesthesiologist in the operating room is a significant challenge that is in urgent need of being addressed. Assistance is required in interpreting the overwhelming stream of physiological data, intelligently extracting key features from these data, and bringing them to the attention of the clinician.

ELIGIBILITY:
Inclusion Criteria:

* Staff anesthesiologist, fellows and 3rd - 5th year residents will be able to participate in this study.
* Subjects willing to provide informed consent.

Exclusion Criteria:

* Inability/failure to provide informed consent.
* Presence of any of the following conditions oPrevious participation in similar experiment oTaken sedative medication within last 24 hours
* Inability/failure to obtain 75% or above in the post-training quiz on the correct use of the eVent.
* Evaluation will be immediately discontinued at request of subject at any point during the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: anesthesiologists, anesthesia residents and fellows
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2010-12; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Ansermino, Principal Investigator — University of British Columbia
Locations (1):
- BC Children's Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Gorges M, Winton P, Koval V, Lim J, Stinson J, Choi PT, Schwarz SK, Dumont GA, Ansermino JM. An evaluation of an expert system for detecting critical events during anesthesia in a human patient simulator: a prospective randomized controlled study. Anesth Analg. 2013 Aug;117(2):380-91. doi: 10.1213/ANE.0b013e3182975b63. Epub 2013 Jun 18. PMID 23780423